CLINICAL TRIAL: NCT04577443
Title: To Investigate the Headache Induction and the Cerebral Hemodynamic Changes After Infusion of Adenosine in Healthy Volunteers and Migraine Patient
Brief Title: The Effect of Adenosine on Cranial Hemodynamic, Headache and Migraine Induction Properties.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Adenosine H-20027630
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Adenosine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adenosine (Active Comparator)
  Interventions: Drug: Adenosine
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Adenosine — To investigate the role of adenosine on cerebral hemodynamic and headache in healthy volunteers and migraine patients
  Arms: Adenosine
Drug: Saline — To investigate the role of saline on cerebral hemodynamic and headache in healthy volunteers and migraine patients
  Arms: Saline

SUMMARY:
Adenosine is a nucleoside that plays a role in both vascular and nociceptive systems, and it has been proposed that adenosine may cause headache in particularly sensitive subjects.

Thus, considerable evidence implied that adenosine plays a role in migraine pathophysiology, it is still unknown if intravenous adenosine infusion provokes migraine attacks in healthy subject or in migraine patients. Furthermore, adenosine's effects on the cerebral hemodynamic remains unknown.

This study aims to clarify a possible coherence between adenosine and headache/migraine. In general, the study will contribute to a greater understanding of migraine pathogenesis and possibly lead to development of specific migraine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients without aura who fulfill criteria in the international classification of headaches. This does not apply to healthy volunteers.
* 18-60 years.
* 50-90 kg.
* Women of childbearing potential must use adequate contraception

Exclusion Criteria:

* Headache less than 48 hours before the tests start
* All primary headaches, except migraine without aura for migraine patients, according to international classification of headache
* Daily consumption of drugs of any kind other than oral contraceptives
* Pregnant or nursing women.
* Cardiovascular disease of any kind, including cerebrovascular diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Occurrence and change of migraine attack | Before (-10 minutes) and after infusion (+12 hours) of adenosine compared with before and after infusion of saline
  Occurrence and of migraine according to international criteria

SECONDARY OUTCOMES:
Change in cerebral hemodynamic | Before (-10 minutes) and after infusion (+12 hours) of adenosine compared with before and after infusion of saline
  Change on velocity of media cerebri artery.
Occurrence and change of headache | Before (-10 minutes) and after infusion (+12 hours) of adenosine compared with before and after infusion of saline
  Occurrence of headache measured by numerical rating scale (NRS)
Change of diameter of the artery | Before (-10 minutes) and after infusion (+12 hours) of adenosine compared with before and after infusion of saline
  Change of diameter of superficial temporal artery and radial artery. The diameter will be measured by millimeter (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Principal Investigator — Danish Headache Center
Locations (1):
- Rigshospitalet-Glostrup, Glostrup Municipality, Nordre Ringvej 57, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thuraiaiyah J, Al-Karagholi MA, Elbahi FA, Zhuang ZA, Ashina M. Adenosine causes short-lasting vasodilation and headache but not migraine attacks in migraine patients: a randomized clinical trial. Pain. 2023 May 1;164(5):1118-1127. doi: 10.1097/j.pain.0000000000002804. Epub 2022 Oct 17. PMID 36251971